CLINICAL TRIAL: NCT05843305
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of BPI-452080 in Subjects With Solid Tumors
Brief Title: A Study of BPI-452080 in Subjects With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTP-661811
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Solid Tumor; Renal Cell Carcinoma; Von Hippel-Lindau Disease
MeSH Terms: conditions — Carcinoma, Renal Cell; von Hippel-Lindau Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Oral tablets taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 21 days in duration with BPI-452080 administered once daily.
  Interventions: Drug: BPI-452080
- Dose Expansion (Experimental): Oral tablets administered at MTD/RP2D defined dose. Each treatment cycle will be 21 days in duration with BPI-452080 administered once daily.
  Cohort 1: Locally Advanced or Metastatic ccRCC Cohort 2: VHL disease associated RCC Cohort 3: Other Advanced Solid Tumors
  Interventions: Drug: BPI-452080

INTERVENTIONS:
Drug: BPI-452080 — Subjects will receive BPI-452080 until disease progression

SUMMARY:
This open-label Phase 1 study will evaluate the efficacy and safety of BPI-452080 in patients with Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic solid tumor patients, who had disease progression after standard therapy, intolerable to standard therapy, refuse to standard therapy or for whom no standard therapy exists
* Dose expansion phase:

Arm1：has locally advanced or metastatic ccRCC and has progressed during treatment with at least one prior therapeutic regimen Arm2：Von Hippel-Lindau Disease-Associated Clear Cell Renal Cell Carcinoma Arm3：Other solid tumors

* Adequate organ function
* Evaluable lesion required for dose escalation phase and at least 1 measurable lesion required for dose expansion phase

Exclusion Criteria:

* Has received prior treatment with another HIF-2α inhibitor
* Inadequate wash-out of prior therapies described per protocol, which may include anti-tumor therapies, tumor adjuvant drugs, organ or stem cell transplantation, moderate or strong CYP3A inhibitor or inducer, etc
* Patients with major surgery within 4 weeks, severe or unstable systemic disease, unstable/symptomatic CNS metastasis, other malignant tumors, ILD, clinical significant cardiac disease, bleeding or embolic disease, active infectious disease, or other medical or psychiatric condition that might interfere with participation in the trial or interfere with the interpretation of trial results, in the opinion of the investigator or medical monitor
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2023-04-28 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
adverse events (AEs) | Through the Phase I, approximately 24 months
  Safety and tolerability will be assessed by monitoring frequency, duration and severity of adverse events

SECONDARY OUTCOMES:
Cmax | Through the Phase I, approximately 24 months
  Maximum observed concentration
Tmax | Through the Phase I, approximately 24 months
  Time to reach maximum observed plasma concentration
t1/2 | Through the Phase I, approximately 24 months
  Half-life time
the objective response rate（ORR） | Through the Phase I, approximately 24 months
  The proportion of patients with complete response (CR) and partial response (PR) in all patients
Progression free survival (PFS) | Through the Phase I, approximately 24 months
  The time from the date of randomization to disease progression (PD) or death, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Ph.D, Principal Investigator — Fudan University; Jian Zhang, Ph.D, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu
  - Zhejiang Cancer Hospital, Hangzhou
  - Hunan Cancer Hospital, Hunan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan